CLINICAL TRIAL: NCT04951479
Title: Geniculate Artery Embolization for Knee Osteoarthritis
Acronym: GAE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anish Ghodadra (Other)
Responsible Party: Sponsor-Investigator, Anish Ghodadra, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY19010266
Record Dates: First submitted 2021-06-28; First posted 2021-07-06 (Actual); Results first posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Gel-Bead Embolization (Experimental): This is the arm undergoing the genicular artery embolization procedure
  Interventions: Device: Gel-Bead embolization

INTERVENTIONS:
Device: Gel-Bead embolization — OptiSphere is FDA approved for the embolization of hypervascular tumors. The product is crosslinked with glutaraldehyde, which improves the mechanical strength of the spheres and provides controlled degradation after implant. The spherical shape provides smooth embolic delivery and even, predictable distribution. In this study the Optispheres will be used for Geniculate artery embolization (GAE) which is a minimally-invasive procedure that has historically been performed for treatment of patients with recurrent knee hemarthrosis. Embolization is a procedure in which material is used to block small blood vessels. Angiogenesis, or growth of new vessels, has been implicated in the initiation and maintenance of joint inflammation. GAE has been applied to patients with moderate osteoarthritis-related pain refractory to maximal medical management with preliminary studies demonstrating a reduction in patient pain.

SUMMARY:
The purpose of this study is to perform a prospective case series to determine efficacy of transcatheter arterial embolization in treating knee osteoarthritis related pain, improving functionality, and reducing opiate usage in patients with mild to moderate knee osteoarthritis who have failed conservative management.

The Gel-Bead embolization particles will be used to perform geniculate artery embolization (GAE) for the purposes of treatment of osteoarthritis-related knee pain.

DETAILED DESCRIPTION:
Management of mild and moderate knee osteoarthritis is curated to each specific patient and their needs, their quality of life, and desired goals. Weight loss is advised for overweight and obese patients. All patients should attempt extended-duration exercise/physical therapy and realignment therapy. If these conservative lifestyle modifications fail to reduce pain, topical and oral non-steroidal anti-inflammatories are indicated. Escalation of care from here is controversial. Some clinicians opt for adjunctive treatments such as intra-articular injection of steroids or viscosupplementation. Unfortunately, pain alleviation from intra-articular steroids is short-lasting and a recent meta-analysis demonstrated no significant difference between intra-articular hyaluronic acid injection and placebo injection. Finally, weak opioids are an option for patients who continue to have pain despite all the aforementioned treatment measures. Joint replacement is reserved for patients with severe osteoarthritis.

Patients who fail conservative, medical management pose a challenge to clinicians. For decades, there have been no interventions available to these patients between the controversial intra-articular hyaluronic acid injection and joint replacement. Interventional radiology (IR) may provide one possible solution. Geniculate artery embolization (GAE) is a minimally-invasive procedure that has historically been performed for patients with recurrent hemarthrosis. It was recently applied to patients with moderate osteoarthritis refractory to maximal medical management. Several studies have been performed and have found that GAE is safe and improves pain.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between ages 18 and 75 with moderate/severe knee pain secondary to primary osteoarthritis. Moderate/severe pain will be defined as pain 30 mm to 100 mm on the Visual Analog Pain Scale (where 0 denotes 'no pain' and 100 mm denotes worst pain imaginable')
2. Grade 1, 2, or 3 osteoarthritis on the Kellgren-Lawrence grading scale on knee x-ray in the last 6 months
3. Pain must be refractory to 3 months of medical management (which may include a combination of oral analgesics, intraarticular steroids, viscosupplementation, opioid therapy, etc)
4. Patients willing and able to consent to the study

Exclusion Criteria:

1. Kidney dysfunction defined as an estimated GFR < 60 mL/min
2. Acute knee injury
3. Current local infection
4. Prior ipsilateral knee replacement surgery
5. Infectious or inflammatory arthritis
6. History of contrast allergy resulting in anaphylaxis
7. INR (International Normalization Ratio) > 1.6
8. Platelets < 50,000
9. Significant atherosclerosis that would limit angiography
10. Active malignancy
11. Active pregnancy
12. Appropriate candidate for knee replacement surgery determined by clinical and physical examination
13. Recent within 3 months, or active cigarette user

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-11-03 (Actual); Primary Completion 2023-10-26 (Actual); Study Completion 2023-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anish Ghodadra, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Shadyside, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Genicular Artery Embolization Arm: This is the single arm of this cohort study. This cohort underwent the GAE procedure.
Period: Overall Study
Arm/Group | Genicular Artery Embolization Arm
Started | 11
Completed | 10
Not Completed | 1
Not completed — Pre-existing Acute Knee Injury | 1

BASELINE CHARACTERISTICS:
Groups:
- Gel-Bead Embolization: Gel-Bead embolization: Gelbead is FDA approved for the embolization of hypervascular tumors. The product is crosslinked with glutaraldehyde, which improves the mechanical strength of the spheres and provides controlled degradation after implant. The spherical shape provides smooth embolic delivery and even, predictable distribution. In this study the Gelbeads will be used for Geniculate artery embolization (GAE) which is a minimally-invasive procedure that has historically been performed for treatment of patients with recurrent knee hemarthrosis. Embolization is a procedure in which material is used to block small blood vessels. Angiogenesis, or growth of new vessels, has been implicated in the initiation and maintenance of joint inflammation. GAE has been applied to patients with moderate osteoarthritis-related pain refractory to maximal medical management with preliminary studies demonstrating a reduction in patient pain.
Arm/Group | Gel-Bead Embolization
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
KOOS Pain Score [Median (Inter-Quartile Range); unit: score on a scale] — The KOOS Pain score runs from 0 (no pain) to 100 (worst pain).
  score on a scale | 42 [38 to 50]

OUTCOME MEASURES:

1. Primary Outcome: Change in KOOS Pain Score
Description: Change in pain score of at least 10 points based on the KOOS Pain questionnaire. The KOOS Pain score runs from 0 (no pain) to 100 (worst pain). The change in KOOS pain score will be the primary outcome measure. Minimum score is 0 and maximum is 100. higher score is better outcome
Time Frame: Baseline and 6 months from treatment
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Genicular Artery Embolization Arm
Number analyzed (Participants) | 10
score on a scale | 33 [22 to 47]
Statistical Analysis 1: Comparison: Genicular Artery Embolization Arm; Paired t-test of KOOS Pain score pre and 6 months post embolization; Test type: Superiority; p = 0.00041, t-test, 2 sided

2. Secondary Outcome: Change in Knee-related Functionality
Description: Average change in the KOOS Function in Sport and Recreation (FSR). The KOOS FSR score runs from 0 (no symptoms) to 100 (worst symptoms).
Time Frame: Baseline and 6 months from treatment
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Genicular Artery Embolization Arm
Number analyzed (Participants) | 10
score on a scale | 39 [15 to 52]
Statistical Analysis 1: Comparison: Genicular Artery Embolization Arm; Test type: Superiority; p = 0.008, t-test, 2 sided

3. Secondary Outcome: Change in KOOS Quality of Life Scale
Description: Average change in in the KOOS Quality of Life Scale (QoL) score. The KOOS QoL score runs from 0 (no symptoms) to 100 (worst symptoms). An increase in this value is considered improvement.
Time Frame: Baseline and 6 months from treatment
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Genicular Artery Embolization Arm
Number analyzed (Participants) | 10
score on a scale | 42 [17 to 50]
Statistical Analysis 1: Comparison: Genicular Artery Embolization Arm; Test type: Superiority; p = 0.001, t-test, 2 sided

4. Secondary Outcome: Change in 30-second Chair Stand Test
Description: Average change in 30-second chair stand test in number of chair stands. An increase in this value is considered improvement.
Time Frame: Baseline and 6 months from treatment
Measure: Median (Inter-Quartile Range); unit: chair stands
Arm/Group | Genicular Artery Embolization Arm
Number analyzed (Participants) | 10
chair stands | 4.5 [2.3 to 10.3]
Statistical Analysis 1: Comparison: Genicular Artery Embolization Arm; Test type: Superiority; p = 0.00797, t-test, 2 sided; paired t-test

5. Secondary Outcome: 6-minute Walk Test
Description: distance walked (meters) in 6 minutes
Time Frame: Baseline and 6 months from treatment
Population: 6 minute walk test was not conducted due to feasibility issues. Protocol was amended to reflect exclusion of 6 minute walk test
Arm/Group | Gel-Bead Embolization
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Genicular Artery Embolization Arm
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 5/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Genicular Artery Embolization Arm (N=10)
Transient Skin Discoloration of the Knee (Skin and subcutaneous tissue disorders) | 3 (3) — Transient blueish discoloration about the knee related to embolization
Allergic Reaction to Toradol (Skin and subcutaneous tissue disorders) | 2 (2) — Skin Rash secondary to PO Toradol given for post-GAE pain
Fever (Infections and infestations) | 1 (1) — Development of fever >100.4 ºF in within the 5 days following GAE

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-04-08): https://cdn.clinicaltrials.gov/large-docs/79/NCT04951479/Prot_SAP_001.pdf